CLINICAL TRIAL: NCT00002089
Title: An Open-Label Study of the Use of Azithromycin in Patients With Symptomatic Disseminated Mycobacterium Avium-Intracellulare Complex (MAC) Infection Failing Current Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 058C; 066-162
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-07

CONDITIONS: Mycobacterium Avium-Intracellulare Infection; HIV Infections
Keywords: Mycobacterium avium-intracellulare Infection; Acquired Immunodeficiency Syndrome; Azithromycin
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Azithromycin

INTERVENTIONS:
Drug: Azithromycin

SUMMARY:
To evaluate the efficacy and safety of azithromycin given chronically for the treatment of Mycobacterium avium (MAC) bacteremia in patients failing or intolerant of current available MAC therapy.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Disseminated MAC as defined by current (within the last month) positive blood, bone marrow, or liver biopsy culture for MAC, and considered symptomatic (fever, night sweats, anorexia, weight loss, fatigue, or malaise).
* At least 2 months of prior treatment with available combination MAC therapy or less than 2 months of such accompanied by unacceptable adverse effects.
* Life expectancy of more than 2 weeks.
* Approval of eligibility from Pfizer Clinical Monitor.
* Consent of parent or guardian if under legal age of consent.

NOTE:

* Patients who have completed acute treatment with azithromycin for MAC in protocol 066-131 or 066-148 will be exempt from inclusion criteria 1 and 2 and can continue therapy through this protocol if their physician feels they have benefitted from prior azithromycin therapy.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Known hypersensitivity or intolerance to macrolide antibiotics.
* Inability to take oral medications or current condition that is likely to interfere with absorption (e.g., gastrectomy).

Concurrent Medication:

Excluded:

* Other MAC therapy instituted during the first 2 months of the study.
* Other investigational drugs, with the exception of those available through a Treatment IND program.

Patients with the following prior conditions are excluded:

History of hypersensitivity or intolerance to azithromycin.

Prior Medication:

Excluded:

* Other investigational drugs within 7 days of enrollment, with the exception of Treatment IND drugs (such as ddC).

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Pfizer Central Research, Groton, Connecticut, United States